CLINICAL TRIAL: NCT04666753
Title: Retrospective Observational Study to Describe the Evolution of SARS-CoV-2 Disease and the Profile of Patients Treated or Not With Imuno TF® and a Combination of Nutraceuticals and Who Have Tested Positive for COVID-19
Brief Title: Retrospective Study of ImmunoFormulation for COVID-19
Status: Completed | Type: Observational
Sponsor: Fagron Iberica S.A.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: IMUNO TF STUDY
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ImmunoFormulation cohort: Patients treated* with IMUNO TF® with a combination of nutraceuticals.
  *Without restrictions on the adjuvant treatment received.
  Interventions: Dietary Supplement: ImmunoFormulation
- Control cohort: Control cohort: patients not treated* with IMUNO TF® with a combination of nutraceuticals.
  *Without restrictions on the adjuvant treatment received.

INTERVENTIONS:
Dietary Supplement: ImmunoFormulation — The ImmunoFormulation consist of: transfer factors (oligo- and polypeptides from porcine spleen, ultrafiltered at <10 kDa - Imuno TF®) 100 mg, 800 mg anti-inflammatory natural blend (Uncaria tomentosa, Endopleura uchi and Haematoccocus pluvialis - MiodesinTM), 60 mg zinc orotate, 48 mg selenium yeast (equivalent to 96 μg of Se), 20,000 IU cholecalciferol, 300 mg ascorbic acid, 480 mg ferulic acid, 90 mg resveratrol, 800 mg spirulina, 560 mg N-acetylcysteine, 610 mg glucosamine sulphate potassium chloride, and 400 mg maltodextrin-stabilized orthosilicic acid (equivalent to 6 mg of Si - SiliciuMax®).
  Groups: ImmunoFormulation cohort

SUMMARY:
Multicentre, retrospective, observational study to describe the course of SARS-CoV-2 disease in patients treated or not with IMUNO TF ® and a combination of nutraceuticals and who have tested positive in a COVID-19 diagnostic test based on the duration of symptoms.

DETAILED DESCRIPTION:
SAMPLE SIZE JUSTIFICATION The primary objective of the study was to describe the course of SARS-CoV-2 disease in patients treated or not with IMUNO TF® and a combination of nutraceuticals and who have tested positive in a COVID-19 diagnostic test based on the duration of symptoms.

Sample size calculation was established according to the ICH guidelines, where it was specified that the number of patients should be sufficient to provide a safe response about the issues raised.

The mean duration of mild/moderate symptoms of COVID-19 was 11.5±5.7 days. A sample of 18 patients would be sufficient to estimate, with a 95% confidence and a precision of +/- 2.8 days, a mean duration of symptoms with a standard deviation of 5.7 days. Assuming a loss of 10% of patients, the sample size was 20 patients. Considering the two groups of patients (treated with IMUNO TF® / not treated with IMUNO TF®), the sample size was 40 patients, 20 patients per group. The calculations were performed with the help of the PASS package, version 2011.

DATA PROCESSING Study data were collected in a CRD and inserted the data in a database specifically designed for the study. The database included internal consistency ranges and rules to ensure data quality control.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older.
2. Patients who give written informed consent to participate in the study.
3. Patients who have consulted their physician for symptoms associated with SARS-CoV-2 infection between March 2020 and May 2020. Patients were included in one cohort or the other based on the treatment received for improvement of COVID-19 symptoms:

   1. IMUNO TF® cohort: patients treated* with IMUNO TF® with a combination of nutraceuticals
   2. Control cohort: patients not treated* with IMUNO TF® with a combination of nutraceuticals *Without restrictions on the adjuvant treatment received.
4. Patients who have tested positive in a diagnostic test for SARS-CoV-2.
5. Patients with onset of COVID-19 symptoms ≥ 5 days prior to diagnosis of SARS-CoV-2.
6. Patients with data in the medical record from the first visit due to disease symptoms until recovery, or at least 1 month of follow-up of symptoms, whichever occurs first.

Exclusion Criteria:

1. Any medical or psychological condition that, in the physician's opinion, could compromise the patient's ability to give informed consent.
2. Patients requiring hospital admission due to the disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: It was planned to collect data from approximately 40 patients who had tested positive in a diagnostic test for SARS-CoV-2: 20 patients who have been treated with IMUNO TF® with a combination of nutraceuticals and 20 patients who have not been treated with the investigational product.
  All patients who met the screening criteria and gave their informed consent to participate were included consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Clinical symptoms duration | 1 month, starting with after start of treatment.
  To describe the course of SARS-CoV-2 disease in patients treated or not with ImmunoFormulation and who have tested positive in a diagnostic test for COVID-19 based on the duration of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Hudson Polonini, PhD, Study Director — Global Innovation Project Manager
Locations (2):
- Spain (2):
  - Clinic Bascoy, Barcelona
  - Clínica Arvila Magna, Barcelona